CLINICAL TRIAL: NCT00500734
Title: Cardiomyopathy Tissue Bank in a Cancer Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID02-359
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Heart Disease
Keywords: Cardiomyopathy; Tissue Bank; Heart Disease; Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Heart Diseases; Cardiomyopathies; Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue collection. This blood may be studied in the future to try to find possible genetic or biochemical markers that may be the cause of CHF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Disease Patients
  Interventions: Procedure: Blood Sample

INTERVENTIONS:
Procedure: Blood Sample — One time blood draw of 2 teaspoons.

SUMMARY:
Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this laboratory research study is to collect and store blood and tissue from patients who have a diagnosis of heart disease and may be at a high risk for the development of heart failure. This blood may be used in the future to identify genes that may play a role in developing congestive heart failure (CHF) from chemotherapy or other sources.

This is an investigational study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
You will have a one time blood draw of 2 teaspoons of blood for use in future research. This blood may be studied in the future to try to find possible genetic or biochemical markers that may be the cause of CHF. Your blood will be drawn either on an outpatient basis or during a routine visit to the hospital. If you already have a central line or an IV placed, the blood will be drawn at these sites to decrease the pain and discomfort of the blood draw. The information obtained in this study will not be put into your medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at high risk for developing Cardiomyopathy or Congestive Heart Failure.
* Patients two months of age and older.

Exclusion Criteria:

* Those that are not willing to sign an informed consent.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with heart disease and that may be at a high risk for the development of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-12-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Patient Demographic Information (age, sex, race) | One time visit.
Identification biological markers predisposing cancer patients to development of chemotherapy-induced congestive heart failure | One time visit for collection of blood and tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Durand, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org